CLINICAL TRIAL: NCT04830553
Title: Exploring the Suitability of Movement and Sound in Couple Therapy: A Proof-of-Concept Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Humboldt-Universität zu Berlin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SONIFY
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music-based couple therapy. (Experimental): Each couple will receive five treatment sessions, including established methods from client-centered and family-systems psychotherapy as well as "Sentire," a technological approach providing immediate sound feedback for physical distance and touch. Duration of the treatment phase: five weeks.
  Interventions: Behavioral: Music-based couple therapy.
- Waiting list. (No Intervention): Each couple will go through an initial waiting period before the treatment phase. Duration of the waiting period: five weeks.

INTERVENTIONS:
Behavioral: Music-based couple therapy. — Each couple will receive five treatment sessions, including established methods from client-centered and family-systems psychotherapy as well as "Sentire," a technological approach providing immediate sound feedback for physical distance and touch. Duration of the treatment phase: five weeks.
  Arms: Music-based couple therapy.

SUMMARY:
The present phase-IIA waiting-list controlled proof-of-concept trial aims to explore the adequacy of immediate sound feedback for physical distance and touch between individuals as a potential means to complement existing methods in couple therapy. The results obtained will determine the design of a subsequent phase-IIB randomized controlled trial.

DETAILED DESCRIPTION:
According to early 20th century psychoanalysis, the "unsaid" becomes apparent in the relationship between patient and therapist, as well as in metaphors and symbols revealed through unintended utterances, imaginative techniques, and dreams. To convey emotions and thoughts, this method relies on the use of spoken language. Likewise, spoken language remains central to the practice of psychotherapy in subsequent decades, as clinicians and researchers sought to translate and transform major claims of psychoanalysis into newer paradigms, the most prominent of them being cognitive-behavioral, client-centered and family-systems psychotherapy. Inspired by somatic psychology and neuroscience evidence, more recent approaches focus on body and movement to target the "unsaid" beyond spoken language. Funded by the German Federal Ministry of Education and Research, the "Sentire" project attempts to provide immediate sound feedback for physical distance and touch between individuals (www.sentire.me). The present phase-IIA waiting-list controlled proof-of-concept trial aims to explore the adequacy of "Sentire" as a potential means to complement existing methods in couple therapy. The results obtained will determine the design of a subsequent phase-IIB randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* In couple relationship for at least six months;
* Living in shared household or close daily contact.

Exclusion Criteria:

* Currently acute episode of any mental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Couples Satisfaction Index, CSI-32. | Change on the CSI-32, as determined by scores on this outcome measure at the beginning, immediately at the end of the five-week treatment phase or five-week waiting-list period, and at 12-month follow-up.
  This self-report questionnaire was conceived to quantify various aspects of a person's satisfaction in a couple relationship on a Likert scale ranging from 0 (very low satisfaction) to 6 (very high satisfaction).

SECONDARY OUTCOMES:
Change in Beck's Depression Inventory, BDI-II. | Change on the BDI-II, as determined by scores on this outcome measure at the beginning, immediately at the end of the five-week treatment phase or five-week waiting-list period, and at 12-month follow-up.
  This self-report measure of depression severity is known for its good psychometric properties, including construct validity and test-retest reliability.
Change in ICD-10 Symptom Rating, ISR. | Change on the ISR, as determined by scores on this outcome measure at the beginning, immediately at the end of the five-week treatment phase or five-week waiting-list period, and at 12-month follow-up.
  This self-report measure based on the ICD-10 criteria of mental disorders serves as a screening instrument for psychological syndromes.

OTHER OUTCOMES:
Childhood Trauma Questionnaire, CTQ. | Beginning of the treatment phase. (Note: This outcome measure is only assessed once prior to the treatment phase.)
  This self-report measure serves as a covariate to determine the relationship between childhood trauma and present issues in a couple relationship.
Positive and Negative Affect Schedule, PANAS. | Change from beginning to end of each couple therapy session (i.e., outcome measure applied before and within 10 minutes after each meeting).
  This self-report measure serves as an indicator of change in emotional arousal within each couple therapy session.
Standortbestimmung. | Change from beginning to end of each couple therapy session (i.e., outcome measure applied before and within 10 minutes after each meeting).
  This self-report measure serves as an indicator of subjective benefit from the treatment experienced within each couple therapy session.
Working Alliance Inventory. | 12-month follow-up. (Note: This outcome measure is only assessed once at the 12-month follow-up.)
  This self-report measure serves as an indicator of therapeutic relationship quality.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Stahl, PhD, Principal Investigator — University Medicine of Greifswald & Medical School Berlin
Locations (1):
- Humboldt-Universität zu Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No